CLINICAL TRIAL: NCT04258202
Title: The Comparison of Ventilator-driven Alveolar Maneuver in Laparoscopic Surgery； Tidal Volume Controlled vs Positive End Expiratory Pressure Controlled Cycling Maneuvers； a Randomized Controlled Study
Brief Title: Ventilator-driven Alveolar Recruitment Maneuver
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SMC2019-11-117-003
Record Dates: First submitted 2020-02-02; First posted 2020-02-06 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-01

CONDITIONS: Postoperative Atelectasis; Ventilator Lung; Atelectasis; Recruitment
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- positive end expiratory pressure group (Experimental): Alveolar recruitment maneuver is performed after intubation, pneumoperitoneum, closure of abdominal fascia. PEEP increased in a stepwise manner from 5 to 20 cmH2O, until plateau pressure 30 cmH2, then 10 breaths. After recruitment, ventilation sets at tidal volume 7 mL/kg with positive end expiratory pressure (PEEP) 5cmH2O.
  Interventions: Other: Alveolar recruitment maneuver
- tidal volume group (Experimental): Alveolar recruitment maneuver is performed after intubation, pneumoperitoneum, closure of abdominal fascia. Tidal volume increased in steps of 4mL/kg of ideal body weight until plateau pressure 30 cmH2O, then 10 breaths. After recruitment, ventilation sets at tidal volume 7 mL/kg with PEEP 5 cmH2O.
  Interventions: Other: Alveolar recruitment maneuver

INTERVENTIONS:
Other: Alveolar recruitment maneuver — The two methods for performing an alveolar recruitment maneuver. Alveolar recruitment maneuvers consisted of a stepwise increase in tidal volume to a plateau pressure of 30 cm H2O versus a stepwise increase in PEEP H2O to a plateau pressure of 30 cm H2O.

SUMMARY:
During laparoscopic surgery, gas infiltration and head down position cause pulmonary atelectasis. Alveolar recruitment maneuvers are beneficial in reopening collapsed alveoli and improving lung mechanics. Ventilator-driven Alveolar recruitment maneuvers may restore lung volume but it remains unknown which method is most effective. The primary aim was to compare the efficacy of two ventilator-driven ARMs method using incremental tidal volume or positive end expiratory pressure(PEEP) until plateau pressure 30 cmH20 (within driving pressure 20 cmH20).

DETAILED DESCRIPTION:
General anesthesia promotes the formation of atelectasis, which negatively impacts respiratory function and may be associated with subsequent pulmonary complications. Especially, during laparoscopic surgery, gas infiltration and head down position cause pulmonary atelectasis. Alveolar recruitment maneuvers are beneficial in reopening collapsed alveoli and improving lung mechanics, suggesting that performing an Alveolar recruitment maneuvers after intubation, circuit disconnection, position change, intraabdominal gas infiltration.

Conventional manual ARM is performed by sustained lung inflation using the reservoir bag on the anaesthesia machine with the adjustable pressure-limiting valve set to the desired inflation pressure. However, the manual ARM can lead to brief loss of positive pressure when switching back to the ventilator circuit, which results in re-collapse of alveoli. For this reason, investigators try to compare the methods of the ventilator-driven ARM.

ELIGIBILITY:
Inclusion Criteria:

* patients who receive laparoscopic surgery in trendelenberg position

Exclusion Criteria:

* Patients who are simultaneously participating in other studies
* Patients who are scheduled to leave the intensive care unit after surgery
* Patients with obstructive or restrictive pattern of Severe or moderate grade on Pulmonary function test
* High risk in cardiovascular events (expected postoperative cardiovascular event > 5%)
* Patients with emphysema confirmed by imaging test
* patients with obesity BMI > 35 kg / m2

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-08 (Actual)

PRIMARY OUTCOMES:
the change of Atelectasis volume | intraoperative time point of intubation, pneumoperitoneum and trendelenberg position, end of surgery
  electrical impedance tomography monitoring: end-expiratory lung impedance, atelectasis (%)

SECONDARY OUTCOMES:
the change of lung compliance value | intraoperative time point of intubation, pneumoperitoneum and trendelenberg position, end of surgery
  comparison of lung compliance mL/cmH2O (static compliance=tidal volume/driving pressure) before/after recruitment maneuver
the change of arterial blood gas analysis | intraoperative time point of intubation, pneumoperitoneum and trendelenberg position, end of surgery
  comparison of PaO2/fraction of inspired oxygen (FiO2) mmHg before/after recruitment maneuver
the change of driving pressure value | intraoperative time point of intubation, pneumoperitoneum and trendelenberg position, end of surgery
  comparison of driving pressure cmH2O (plateau pressure-positive end expiratory pressure) before/after recruitment maneuver
the change of peak pressure value | intraoperative time point of intubation, pneumoperitoneum and trendelenberg position, end of surgery
  comparison peak pressure (cmH2O) before/after recruitment maneuver
The difference of atelectasis | at postoperative 30 minutes
  atelectasis score by lung ultrasonography (score range 0~36)

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung medical center, Seoul, South Korea